CLINICAL TRIAL: NCT07193602
Title: Home-based Virtual Reality (VR) Headset-based Dexterity Training in Multiple Sclerosis: a Randomized-controlled Trial
Brief Title: VR-based Dexterity Training in MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Kamm (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Christian Kamm, Prof. Dr. med., Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUKSKAMM003
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Headset-based dexterity training; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized-controlled, home-based, multi-center, rater-blinded parallel-arm pilot study.
Who Masked: Outcomes Assessor
Masking Description: Raters will not be involved in the screening and randomisation process and blinded with regard to the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental intervention = training intervention (Group1) (Experimental): Eight training programs will be performed addressing different key movements of the hand/arm. All training programs will be performed in sitting position. Training will be performed for 4 weeks, 5 days/week. All 8 training programs will be performed on every training day which corresponds to approximately 20min training/day.
  Interventions: Device: VR-based dexterity training in MS
- Control inervention = Sham-Intervention (Group2) (Sham Comparator): The Sham-Intervention will be the commercially available meditations App "Tripp®". During a period of four weeks, patients will perform the Sham intervention 3 times a week, each session being approximately 20 minutes.
  Interventions: Other: mediation program

INTERVENTIONS:
Device: VR-based dexterity training in MS — Training of limited manual dexterity in people with multiple sclerosis through a specially developed home-based dexterity training programm using a virtual headset
  Arms: Experimental intervention = training intervention (Group1)
Other: mediation program — Sham Training is the comparator. The Sham group is performing a commercially available mediation programm TRIPP:
  Arms: Control inervention = Sham-Intervention (Group2)

SUMMARY:
The aim of the study is to investigate if a specifically developed home-based dexterity training intervention using a Virtual Reality (VR) Headset (Meta quest 2) improves impaired manual dexterity in persons with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* MS patients with relapsing-remitting MS (RRMS), secondary-progressive MS (SPMS) or primary progressive MS (PPMS) according to the revised McDonald's criteria (Thompson et al. 2017).

Age between 18 and 75 years.

Written informed consent signed by the subject must be obtained prior to study start

Patient must complain about MS related impaired manual dexterity negatively affecting ADL and/or QoL.

Patients must have a pathological 9-Hole-Peg-Test (9HPT) as defined by Oxford Grice et al. 2003.

Patients must have Arm function in multiple sclerosis questionnaire (AMSQ) score >41

Exclusion Criteria:

* A relapse that started within 60 days prior to screening.

Rapidly progressive disease.

Any disease/condition that impaired manual dexterity besides MS

Any disease other than MS that could possibly explain the patient's signs and symptoms

Medical or psychiatric conditions that compromise the ability to comply with the protocol, or to complete the study

A history of drug abuse in the 12 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Arm Function Score in Multiple Sclerosis Questionnaire | 4 weeks
  The Arm Function in Multiple Sclerosis Questionnaire (AMSQ) measures manual dexterity in patients with MS. It contains 31 questions on a unidimensional scale. One final sum score is obtained with higher scores indicating more dexterous difficulties.

SECONDARY OUTCOMES:
Time for completing the Nine-hole-Peg-Test (9HPT) | 4 weeks
  The Nine-hole-Peg-Test (9HPT) is reliable (ICC values 0.80-0.99), valid and sensitive in detecting impaired dexterity in patients with MS. Patients were seated at a table with a shallow container holding nine pegs and a plastic block with nine empty holes. All pegs had to be put one at a time into the holes and then removed again one at a time into the shallow container. The time to complete the task was recorded twice on both hands and mean values were taken for each hand.
Time for completion the Coin rotation task (CRT) | 4 Weeks
  The Coin rotation task (CRT) has been validated in assessing manual dexterity in patients with MS . Patients had to rotate a 50 Swiss Rappen coin (corresponding to a dime or 2-cent Euro coin) as fast as possible between their thumb, index and middle finger. The time to perform 20 half turns was measured twice on both hands and mean values were taken for each hand.
The highest strength value resulting from the Handheld JAMAR dynamometer | 4 Weeks
  The Handheld JAMAR dynamometer is a reliable (ICC values 0.85 - 0.98) and valid test to measures isometric grip strength of the hands in healthy subjects and in MS patients. It is performed in an upright seating position with 90° flexion of the elbow next to the body. The highest value (kilograms force) of two maximum voluntary grip strength movements was taken for each hand.
Value resulting from the Multiple Sclerosis Impact Scale 29 (MSIS 29) | 4 Weeks
  The Multiple Sclerosis Impact Scale 29 (MSIS 29) is valid and reliable in measuring the impact of MS on ADL. It contains 29 items comprising to a physical (MSIS-29 physical) and psychological impact scale (MSIS-29 psychological). All items are scored from 'not at all' to 'extremely' on a five-point Likert scale.
Scores of eEDSS | 4 Weeks
  Comparing the subscores of the upper extremity

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - MS Centre, Neurology, University hospital Basel, Basel, Basel
  - Lucerne Cantonal Hospital, Lucerne, Canton of Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yancosek KE, Howell D. A narrative review of dexterity assessments. J Hand Ther. 2009 Jul-Sep;22(3):258-69; quiz 270. doi: 10.1016/j.jht.2008.11.004. Epub 2009 Feb 12. PMID 19217254
- [Background] Winberg C, Kylberg M, Pettersson C, Harnett T, Hedvall PO, Mattsson T, Mansson Lexell E. The Use of Apps for Health in Persons with Multiple Sclerosis, Parkinson's Disease and Stroke - Barriers and Facilitators. Stud Health Technol Inform. 2017;242:638-641. PMID 28873864
- [Background] Vanbellingen T, van Beek J, Nyffeler T, Urwyler P, Nef T, Bohlhalter S. Tablet app-based dexterity-training in patients with Parkinson's disease: Pilot feasibility study. Ann Phys Rehabil Med. 2021 Jul;64(4):101419. doi: 10.1016/j.rehab.2020.06.004. Epub 2020 Oct 6. No abstract available. PMID 32755640
- [Background] van Beek JJW, van Wegen EEH, Rietberg MB, Nyffeler T, Bohlhalter S, Kamm CP, Nef T, Vanbellingen T. Feasibility of a Home-Based Tablet App for Dexterity Training in Multiple Sclerosis: Usability Study. JMIR Mhealth Uhealth. 2020 Jun 9;8(6):e18204. doi: 10.2196/18204. PMID 32515747
- [Background] van Beek JJW, van Wegen EEH, Bol CD, Rietberg MB, Kamm CP, Vanbellingen T. Tablet App Based Dexterity Training in Multiple Sclerosis (TAD-MS): Research Protocol of a Randomized Controlled Trial. Front Neurol. 2019 Feb 11;10:61. doi: 10.3389/fneur.2019.00061. eCollection 2019. PMID 30804879
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Thirumalai M, Rimmer JH, Johnson G, Wilroy J, Young HJ, Mehta T, Lai B. TEAMS (Tele-Exercise and Multiple Sclerosis), a Tailored Telerehabilitation mHealth App: Participant-Centered Development and Usability Study. JMIR Mhealth Uhealth. 2018 May 24;6(5):e10181. doi: 10.2196/10181. PMID 29798832
- [Background] Tacchino A, Pedulla L, Bonzano L, Vassallo C, Battaglia MA, Mancardi G, Bove M, Brichetto G. A New App for At-Home Cognitive Training: Description and Pilot Testing on Patients with Multiple Sclerosis. JMIR Mhealth Uhealth. 2015 Aug 31;3(3):e85. doi: 10.2196/mhealth.4269. PMID 26323749
- [Background] Steinheimer S, Wendel M, Vanbellingen T, Westers LT, Hodak J, Blatter V, Uitdehaag BMJ, Kamm CP. The Arm Function in Multiple Sclerosis Questionnaire was successfully translated to German. J Hand Ther. 2018 Jan-Mar;31(1):137-140.e1. doi: 10.1016/j.jht.2017.09.010. No abstract available. PMID 29102479
- [Background] Riazi A, Hobart JC, Lamping DL, Fitzpatrick R, Thompson AJ. Multiple Sclerosis Impact Scale (MSIS-29): reliability and validity in hospital based samples. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):701-4. doi: 10.1136/jnnp.73.6.701. PMID 12438473
- [Background] Peolsson A, Hedlund R, Oberg B. Intra- and inter-tester reliability and reference values for hand strength. J Rehabil Med. 2001 Jan;33(1):36-41. doi: 10.1080/165019701300006524. PMID 11480468
- [Background] Paltamaa J, West H, Sarasoja T, Wikstrom J, Malkia E. Reliability of physical functioning measures in ambulatory subjects with MS. Physiother Res Int. 2005;10(2):93-109. doi: 10.1002/pri.30. PMID 16146327
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] McGuigan C, Hutchinson M. The multiple sclerosis impact scale (MSIS-29) is a reliable and sensitive measure. J Neurol Neurosurg Psychiatry. 2004 Feb;75(2):266-9. PMID 14742602
- [Background] Marrie RA, Leung S, Tyry T, Cutter GR, Fox R, Salter A. Use of eHealth and mHealth technology by persons with multiple sclerosis. Mult Scler Relat Disord. 2019 Jan;27:13-19. doi: 10.1016/j.msard.2018.09.036. Epub 2018 Oct 2. PMID 30296732
- [Background] Mokkink LB, Knol DL, van der Linden FH, Sonder JM, D'hooghe M, Uitdehaag BMJ. The Arm Function in Multiple Sclerosis Questionnaire (AMSQ): development and validation of a new tool using IRT methods. Disabil Rehabil. 2015 Dec;37(26):2445-2451. doi: 10.3109/09638288.2015.1027005. Epub 2015 Mar 24. PMID 25801923
- [Background] Lamers I, Kelchtermans S, Baert I, Feys P. Upper limb assessment in multiple sclerosis: a systematic review of outcome measures and their psychometric properties. Arch Phys Med Rehabil. 2014 Jun;95(6):1184-200. doi: 10.1016/j.apmr.2014.02.023. Epub 2014 Mar 13. PMID 24631802
- [Background] Kamm CP, Uitdehaag BM, Polman CH. Multiple sclerosis: current knowledge and future outlook. Eur Neurol. 2014;72(3-4):132-41. doi: 10.1159/000360528. Epub 2014 Jul 30. PMID 25095894
- [Background] Kamm CP, Mattle HP, Muri RM, Heldner MR, Blatter V, Bartlome S, Luthy J, Imboden D, Pedrazzini G, Bohlhalter S, Hilfiker R, Vanbellingen T. Home-based training to improve manual dexterity in patients with multiple sclerosis: A randomized controlled trial. Mult Scler. 2015 Oct;21(12):1546-56. doi: 10.1177/1352458514565959. Epub 2015 Jan 26. PMID 25623246
- [Background] Kamm CP, Blattler R, Kueng R, Vanbellingen T. Feasibility and usability of a new home-based immersive virtual reality headset-based dexterity training in multiple sclerosis. Mult Scler Relat Disord. 2023 Mar;71:104525. doi: 10.1016/j.msard.2023.104525. Epub 2023 Jan 20. PMID 36738693
- [Background] Kamm CP, Kueng R, Blattler R. Development of a new immersive virtual reality (VR) headset-based dexterity training for patients with multiple sclerosis: Clinical and technical aspects. Technol Health Care. 2024;32(2):1067-1078. doi: 10.3233/THC-230541. PMID 37545286
- [Background] Kalkers NF, Galan I, Kerbrat A, Tacchino A, Kamm CP, O'Connell K, McGuigan C, Edan G, Montalban X, Uitdehaag BM, Mokkink LB. Differential item functioning of the Arm function in Multiple Sclerosis Questionnaire (AMSQ) by language, a study in six countries. Mult Scler. 2021 Jan;27(1):90-96. doi: 10.1177/1352458519895450. Epub 2019 Dec 17. PMID 31845614
- [Background] Jonsdottir J, Perini G, Ascolese A, Bowman T, Montesano A, Lawo M, Bertoni R. Unilateral arm rehabilitation for persons with multiple sclerosis using serious games in a virtual reality approach: Bilateral treatment effect? Mult Scler Relat Disord. 2019 Oct;35:76-82. doi: 10.1016/j.msard.2019.07.010. Epub 2019 Jul 20. PMID 31352180
- [Background] Johansson S, Ytterberg C, Claesson IM, Lindberg J, Hillert J, Andersson M, Widen Holmqvist L, von Koch L. High concurrent presence of disability in multiple sclerosis. Associations with perceived health. J Neurol. 2007 Jun;254(6):767-73. doi: 10.1007/s00415-006-0431-5. Epub 2007 Apr 2. PMID 17401746
- [Background] Hollywood RA, Poyade M, Paul L, Webster A. Proof of Concept for the Use of Immersive Virtual Reality in Upper Limb Rehabilitation of Multiple Sclerosis Patients. Adv Exp Med Biol. 2022;1356:73-93. doi: 10.1007/978-3-030-87779-8_4. PMID 35146618
- [Background] Hobart J, Lamping D, Fitzpatrick R, Riazi A, Thompson A. The Multiple Sclerosis Impact Scale (MSIS-29): a new patient-based outcome measure. Brain. 2001 May;124(Pt 5):962-73. doi: 10.1093/brain/124.5.962. PMID 11335698
- [Background] Heldner MR, Vanbellingen T, Bohlhalter S, Mattle HP, Muri RM, Kamm CP. Coin rotation task: a valid test for manual dexterity in multiple sclerosis. Phys Ther. 2014 Nov;94(11):1644-51. doi: 10.2522/ptj.20130252. Epub 2014 Jun 19. PMID 24947199
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] D'Souza M, Heikkila A, Lorscheider J, Haller V, Kravalis K, Gysin S, Fuertes NAC, Fricker E, Lam E, Higgins P, Tomic D, Papadopoulou A, Kappos L. Electronic Neurostatus-EDSS increases the quality of expanded disability status scale assessments: Experience from two phase 3 clinical trials. Mult Scler. 2020 Jul;26(8):993-996. doi: 10.1177/1352458519845108. Epub 2019 May 7. PMID 31060429
- [Background] Bertoni R, Mestanza Mattos FG, Porta M, Arippa F, Cocco E, Pau M, Cattaneo D. Effects of immersive virtual reality on upper limb function in subjects with multiple sclerosis: A cross-over study. Mult Scler Relat Disord. 2022 Sep;65:104004. doi: 10.1016/j.msard.2022.104004. Epub 2022 Jun 30. PMID 35797804